CLINICAL TRIAL: NCT02323360
Title: A Randomised Phase III Trial on Stereotactic Body Radiotherapy (SBRT) After Incomplete Transcatheter Arterial Embolization (TAE) or Chemoembolization (TACE) Versus Exclusive TAE or TACE for Inoperable Hepatocellular Carcinoma (HCC)
Brief Title: A Trial on SBRT After Incomplete TAE or TACE Versus Exclusive TAE or TACE For Treatment of Inoperable HCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too slow enrollment
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1315
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: SBRT; TACE; TAE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stereotactic body radiation therapy (Experimental): HCC after incomplete TAE or TACE treated by SBRT
  Interventions: Radiation: SBRT
- TACE/TAE (Active Comparator): HCC after incomplete TAE or TACE treated by a new cycle of TAE or TACE
  Interventions: Procedure: TACE

INTERVENTIONS:
Radiation: SBRT — Patients with single nodule no more 5 cm or 1- 3 nodules no more 3 cm in diameter after incomplete TAE or TACE, are randomized to stereotactic radiotherapy in 3 or 6 daily fractions
  Other Names: Stereotactic body radiation therapy
  Arms: Stereotactic body radiation therapy
Procedure: TACE — Patients with single nodule no more 5 cm or 1- 3 nodules no more 3 cm in diameter after incomplete TAE or TACE, are randomized to a new cycle of TAE or TACE
  Other Names: Transcatheter arterial chemoembolization
  Arms: TACE/TAE

SUMMARY:
The trial is a multicentre, prospective, randomised controlled, unblinded, parallel-group superiority trial of SBRT versus standard TAE/TACE for the curative treatment of inoperable HCC treated with a TAE/TACE incomplete cycle.

DETAILED DESCRIPTION:
In this phase III study patients with inoperable HCC single nodule no more 5 cm or 1- 3 nodules no more 3 cm in diameter after incomplete TAE or TACE, are randomized to stereotactic radiotherapy in 3 or 6 daily fractions or to a new cycle of TAE or TACE. A total of 80 patients (40 in each arm) will be recruited into the trial over a 2 years period and will be randomised on an equal basis to either SBRT or TAE/TACE. The follow-up period will be finished 1.5 years after the final patient is randomised.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Karnofsky index >70%
* Child-Turgotte-Pugh A or B liver score.
* An initial diagnosis of primary HCC or recurrence.
* A technically unresectable lesion or medically contraindicated surgery or a case in which surgery was declined.
* HCC (single nodule ≤ 5 cm or max 3 nodules ≤ 3 cm) diagnosed by histology or non-invasive EASL criteria
* Baseline CT or MRI and bone scan without evidence of radiologically definable major vascular invasion or extrahepatic disease
* Hb >10.5.0 g/%, WBC >3.000 cells/mm3, platelets >50.000 cells/mm3, bilirubin <2 mg/dl, aspartate and alanine aminotransferase levels <5 times upper normal limit, and prothrombin time-international normalized ratio ≤ 2;
* Serum creatinine <1.7 mg/dl
* Previously incomplete TAE or TACE with radiologically defined residual disease.
* Informed consent

Exclusion Criteria:

* Extrahepatic disease and refractory ascites.
* Previous abdominal radiation therapy (RT)
* Hemorrhage/bleeding event = Grade 3 within 4 weeks of enrollment in the study.
* Pregnant or breastfeeding patients.
* Patients with uncontrolled infections or HIV seropositive patients.
* Mental conditions rendering the patient incapable to understand the nature, scope, and consequences of the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Local control (efficacy of SBRT in selected HCC patients with an incomplete response after TACE/TAE) | 1.5 years
  This is a study designed to evaluate the efficacy of SBRT in selected HCC patients with an incomplete response after TACE/TAE.

SECONDARY OUTCOMES:
progression free-survival | 1.5 years
overall survival | 1.5 years
toxicity (incidence of acute and late complications) | 1.5 years
  incidence of acute and late complications

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Derived] Comito T, Loi M, Franzese C, Clerici E, Franceschini D, Badalamenti M, Teriaca MA, Rimassa L, Pedicini V, Poretti D, Solbiati LA, Torzilli G, Ceriani R, Lleo A, Aghemo A, Santoro A, Scorsetti M. Stereotactic Radiotherapy after Incomplete Transarterial (Chemo-) Embolization (TAE\TACE) versus Exclusive TAE or TACE for Treatment of Inoperable HCC: A Phase III Trial (NCT02323360). Curr Oncol. 2022 Nov 16;29(11):8802-8813. doi: 10.3390/curroncol29110692. PMID 36421345